CLINICAL TRIAL: NCT01118312
Title: Study of Asthma and Nasal Steroids for the American Lung Association-Airways Clinical Research Centers
Brief Title: Study of Asthma and Nasal Steroids
Acronym: STAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALAACRC-11; R01 HL089464-01A2 (Other: NIH/NHLBI); R01 HL00895101-01A2 (Other: NIH/NHLBI)
Record Dates: First submitted 2010-04-28; First posted 2010-05-06 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Asthma; Rhinitis; Sinusitis
Keywords: Asthma; Rhinitis; Sinusitis; Chronic; ACRC; STAN; Nasal steroid; Mometasone; Nasal spray
MeSH Terms: conditions — Asthma; Rhinitis; Sinusitis; Bronchiolitis Obliterans Syndrome | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal Steroid (Active Comparator): Intranasal mometasone, 1 spray (age < 12 yr) or 2 sprays (age >= 12 yrs) each nostril once a day
  Interventions: Drug: Mometasone Furoate monohydrate
- Placebo (Placebo Comparator): Intranasal placebo, 1 spray (age < 12 yr) or 2 sprays (age >= 12 yrs) each nostril once a day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate monohydrate — Intranasal mometasone, 1 spray (age < 12 yr) or 2 sprays (age >= 12 yrs) each nostril once a day for 6 months
  Other Names: Nasonex
  Arms: Nasal Steroid
Other: Placebo — Intranasal placebo spray
  Arms: Placebo

SUMMARY:
The trial will study the effectiveness of nasal steroids for the treatment of chronic rhinitis and/or sinusitis on asthma control.

DETAILED DESCRIPTION:
Previous trials completed by the American Lung Association-Airways Clinical Research Centers (ALA-ACRC) network have identified rhinitis and/or sinusitis as a significant co-morbidity in people with asthma that affects asthma symptoms and control. The objective of this clinical trial is to determine if treatment of chronic rhinitis and/or sinusitis with nasal steroids improves control of asthma in children and adults. Although chronic rhinitis and/or sinusitis have been associated with poor asthma control and increased health care utilization, the effect of treating these diseases on asthma control is not known. This will be a six-month randomized, double-blinded, placebo-controlled trial enrolling 380 participants, 190 children and 190 adults, with poorly controlled asthma and chronic rhinitis/sinusitis. Participants will be randomized to receive nasal steroid or a matching placebo in addition to their regular asthma treatments. The primary objective of the trial will be to evaluate whether the addition of treatment with nasal steroids improves asthma control. We will perform allergy skin testing on all participants and keep a record of pollen counts at all centers, to determine if allergy is an important factor in the response to nasal steroid in participants.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma
* At least 12% increase in forced expiratory volume at one second (FEV1) after 2-4 puffs of albuterol or positive methacholine challenge (20% fall in FEV1 at less than 16 mg/ml methacholine); either of these can be available from the last 2 years before enrollment
* Poorly controlled asthma as documented by a score of 19 or less on the Asthma Control Test (ACT) for participants 12 and older, and a Childhood Asthma Control Test (C-ACT) for 6-11 years(both V1 and V2).
* Chronic symptoms of rhinitis and sinusitis as measured by a mean score of 1 on the Sino-nasal questionnaire
* Males and females, age 6 and older

Exclusion Criteria:

* Co-morbidity that predisposes to complicated rhino-sinusitis (e.g., cystic fibrosis, insulin dependent diabetes mellitus, immunodeficiency disorder)
* Chronic diseases (other than asthma) that in the opinion of the investigator would prevent participation in the trial or put the participant at risk by participation, e.g. chronic diseases of the lung (other than asthma), heart, liver, kidney or nervous system.
* History of sinus surgery in last 6 months
* Systemic/nasal steroids within last 4 weeks
* Anti-leukotriene medication
* History of upper airway symptoms for less than 8 weeks at the time of enrollment
* Fever > 38.3 degrees Celsius or patient history of fever in last 10 days
* Greater than 10 pack year smoking history or active smoking within the last 6 months
* FEV1 < 50% predicted
* Females of childbearing potential that are pregnant or lactating, or unwilling to practice an adequate birth control method
* Allergy or intolerance to nasal mometasone
* Cataracts, history of glaucoma, or other conditions resulting in increased intraocular pressure
* Any investigational drug in the last 6 weeks
* Inability to comply with study procedures, including:

  * Inability or unwillingness to provide informed consent (or assent in the case of a minor)
  * Inability to take study medication
  * Inability to perform baseline measurements
  * Completion of less than 10 of the 14 days of screening period diary entry
  * Inability to be contacted by phone
  * Intention to move out of the area within 6 months

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dixon, MD, Principal Investigator — University of Vermont
Locations (19):
- United States (19):
  - University of Arizona, Tucson, Arizona
  - University of California, San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - Univeristy of Miami School of Medicine, Miami, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - University of Missouri, Kansas City School of Medicine, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - North Shore-Long Island Jewish Health System, New Hyde Park, New York
  - New York University School of Medicine, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Vermont Lung Center at the University of Vermont, Burlington, Vermont
  - Univeristy of Virginia, Charlottesville, Virginia

REFERENCES:
- See also: ALA-ACRC Webpage — http://www.cctrials.org/alaacrc

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Steroid | Placebo
Started | 189 | 199
Completed | 155 | 164
Not Completed | 34 | 35
Not completed — Lost to Follow-up | 33 | 32
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Steroid | Placebo | Total
Number analyzed (Participants) | 189 | 199 | 388
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72 | 79 | 151
  Between 18 and 65 years | 117 | 120 | 237
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 106 | 211
  Male | 84 | 93 | 177

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Test (ACT)
Description: Asthma Control Test for adults (score range: 5-25); higher score indicates better asthma control
Time Frame: 24 weeks
Population: Analysis of adult (18 and above) Asthma Control Scores
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nasal Steroid | Placebo
Number analyzed (Participants) | 117 | 120
units on a scale | 2.95 (0.31) | 2.44 (0.38)

2. Secondary Outcome: Childhood Asthma Control Test
Description: Childhood Asthma Control Test (score range: 0-27); higher score indicates better asthma control
Time Frame: 24 weeks
Population: Analysis of Children (less than 18 years old) Childhood Asthma Control Test scores
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nasal Steroid | Placebo
Number analyzed (Participants) | 72 | 79
units on a scale | 4.15 (0.64) | 4.53 (0.65)

ADVERSE EVENTS:
Arm/Group | Nasal Steroid | Placebo
Serious Adverse Events (participants affected / at risk) | 2/189 | 9/199
Other Adverse Events (participants affected / at risk) | 105/179 | 127/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nasal Steroid (N=189) | Placebo (N=199)
Depression (hospitalized) (Psychiatric disorders) | 1 | 1
Anaphylactic reaction (General disorders) | 1 | 0
Dental abscess (General disorders) | 0 | 1
Headache and high blood pressure (Vascular disorders) | 0 | 1
Dehydration (General disorders) | 0 | 1
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
pneumonia (Infections and infestations) | 0 | 1
Fungus ball of the sinus requiring surgery (Surgical and medical procedures) | 0 | 1
appendicitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nasal Steroid (N=179) | Placebo (N=187)
Headache (Vascular disorders) | 45/140 | 56/148 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Sore throat (General disorders) | 22/174 | 34/175 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Nasal bleed (General disorders) | 10/176 | 15/184 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Nasal pain (General disorders) | 25/162 | 44/168 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Rash (Skin and subcutaneous tissue disorders) | 7/172 | 18/180 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Itching (Skin and subcutaneous tissue disorders) | 17/157 | 23/165 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Dizzy (Ear and labyrinth disorders) | 9/172 | 17/181 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Upper respiratory tract infection (Infections and infestations) | 27/178 | 28/184 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Trouble breathing (Respiratory, thoracic and mediastinal disorders) | 42/136 | 55/152 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Swelling (General disorders) | 10/175 | 19/183 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Cough (Respiratory, thoracic and mediastinal disorders) | 39/133 | 44/157 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.
Dysmenorrhea (Reproductive system and breast disorders) | 10/116 | 14/112 — Counts include the number of individuals who experienced a moderate or severe symptom at follow up. Individuals who had the symptom (moderate or severe) at baseline are excluded as are those with no follow-up data on the adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No